CLINICAL TRIAL: NCT00227318
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Long-term Trial of Preventing Hypertension Using Candesartan Cilexetil 16 mg in Patients With High Normal Blood Pressure (TROPHY)
Brief Title: TROPHY - Candesartan Cilexetil Long-term Hypertension Prevention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: SH-AHM-0030; D2455L00010 (Other: AstraZeneca)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

INTERVENTIONS:
Drug: ATACAND

SUMMARY:
The purpose of this study is to determine the effectiveness of candesartan cilexetil in preventing hypertension in people with high normal blood pressure. Patients will be randomized to either Candesartan or placebo for an initial 2-year period followed by a second 2-year period of placebo for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 30 and 65 (inclusive) at the time of the informed consent process
* have an average clinic BP in the high normal range of < 139/85-89 mmHg or 130-139/< 89 mm Hg (high normal BP range) (mean systolic and/or diastolic pressure based on 3 consecutive measurements) derived from the average of clinic visits 1,2 and 3.

Exclusion Criteria:

* Have proteinuria >1 + (by dipstick method)
* have a stroke, myocardial infarction (MI), transient ischemic attack (TIA), the presence of any clinically significant evidence of atherosclerosis or hypertensive target organ involvement or any significant medical condition that may compromise participation in this study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 1998-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To determine whether candesartan cilexetil 16 mg compared to placebo reduces the crude incidence of hypertension in a population with high normal BP evaluated after a 4-year study period consisting of 2 years of double-blind treatment followed by 2 years

SECONDARY OUTCOMES:
To evaluate the reduction in BP after 2 years treatment with candesartan cilexetil 16 mg vs placebo in patients with high normal BP.
To evaluate the incidence of hypertension after 2 years treatment with candesartan cilexetil 16 mg vs placebo in patients with high normal BP.
To evaluate Health-related Quality of Life yearly during 2 years treatment with candesartan cilexetil 16mg vs placebo and yearly during a 2-year follow up period in patients with high normal BP.

CONTACTS AND LOCATIONS:
Overall Officials: Atacand Medical Science Director, MD, Study Director — AstraZeneca
Locations (42):
- United States (42):
  - Research Site, Mobile, Alabama
  - Research Site, Long Beach, California
  - Research Site, Redondo Beach, California
  - Research Site, Santa Ana, California
  - Research Site, Tustin, California
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bay Pines, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Chelsea, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Florissant, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, Rochester, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Allentown, Pennsylvania
  - Research Site, Fleetwood, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Julius S, Nesbitt SD, Egan BM, Weber MA, Michelson EL, Kaciroti N, Black HR, Grimm RH Jr, Messerli FH, Oparil S, Schork MA; Trial of Preventing Hypertension (TROPHY) Study Investigators. Feasibility of treating prehypertension with an angiotensin-receptor blocker. N Engl J Med. 2006 Apr 20;354(16):1685-97. doi: 10.1056/NEJMoa060838. Epub 2006 Mar 14. PMID 16537662
- [Derived] Kang S, Little RJ, Kaciroti N. Missing not at random models for masked clinical trials with dropouts. Clin Trials. 2015 Apr;12(2):139-48. doi: 10.1177/1740774514566662. Epub 2015 Jan 27. PMID 25627429